CLINICAL TRIAL: NCT03126487
Title: High Intensity Focused Ultrasound Guided by MRI as Thermic Destruction in Primitive Small Size Breast Cancer. Phase II Pilot Study : Effectiveness and Procedures Standardization
Brief Title: High Intensity Focused Ultrasound Guided by MRI as Thermic Destruction in Primitive Small Size Breast Cancer
Acronym: MRHEATBREAST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study do not start due to concurrential trial
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/36
Record Dates: First submitted 2017-04-12; First posted 2017-04-24 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIGH INTENSITY FOCUSED ULTRASOUND (Experimental): HIGH INTENSITY FOCUSED ULTRASOUND
  Interventions: Procedure: HIGH INTENSITY FOCUSED ULTRASOUND

INTERVENTIONS:
Procedure: HIGH INTENSITY FOCUSED ULTRASOUND — HIGH INTENSITY FOCUSED ULTRASOUND GUIDED BY MRI AS THERMIC DESTRUCTION

SUMMARY:
This is a non-randomized, prospective phase II trial evaluating an innovative treatment, focused MRI-guided ultrasound, as thermic destruction in primitive small size breast cancer.

DETAILED DESCRIPTION:
Conservative Breast Treatment (BCT) :

The reference treatment for patients with stage T1 breast cancer is a partial mastectomy followed by radiotherapy (breast). This is a conservative treatment (BCT). Indeed, the survival results of this combined treatment are equivalent to those observed after a total mastectomy alone and is an aesthetically and psychologically more acceptable proposition for patients.

Adjuvant radiotherapy is an essential component of the success of conservative therapy most likely due to the impossibility of surgical treatment of removing all microscopically viable cancer cells. Indeed, in the absence of radiotherapy, partial mastectomy shows a local recurrence rate of 20-40% in case of N0 and 25-50% in case of N + on long-term follow-up data.

The results of the literature are very variable according to the length of the follow-up and the population studied but the adjuvant radiotherapy clearly allows to increase the rate of local control.

It reduces local recurrences to 10% at 12 years in the case of radiotherapy in the breast and 6% in case of boost on the tumor area.

The high sensitivity of breast MRI and emerging issues. The development of breast MRI revealed the incidental discovery of 10 to 40% of additional breast cancer in patients initially explored by mammography and ultrasound standards. These cancers discovered at early stages and of small size complicate the strategy of local management and incite to develop techniques alternative to the surgery.

Several minimally invasive treatments for the local treatment of breast cancers are being studied: BLES (Breast Lesion Excision Sample), cryotherapy, radiofrequency, laser and microwaves. Among them, focused ultrasound offers a completely non-invasive heat ablation technique.

High intensity focused ultrasound (FUS) and magnetic resonance imaging (MRI) guidance = FUS-MRI High intensity focused ultrasound thermal ablation is an attractive treatment modality for solid tumors because it does not require incision. Moreover, coupled with magnetic resonance, it offers precise targeting and control destruction.

An ablation procedure begins with the acquisition of a series of MRI images centered on the organ to be treated. The radiologist loads the images onto the processing machine and identifies the target volume to be destroyed by segmenting it from the MRI images. The console provides a treatment plan with the necessary parameters to efficiently process the defined region.

High intensity focussed ultrasonic destruction is possible due to the elevation of temperature at the focal point. By analogy, one can compare the technique to the use of a magnifying glass to focus the sun's rays and trigger a flame. In ultrasound diagnostic ultrasound is used without convergence of beams. In the therapeutic application, it is the focusing at a point and the use of high intensities which make it possible to deliver energy in the form of heat. This step is called "sonication". Sonication heats the tissue between 65 and 85 ° C in the well-defined region of the focal point and causes tissue thermo-coagulation.

MRI images acquired during heating allow real-time monitoring of the rise in temperature. This makes it possible to check the position of the sonication and the size of the zone thus coagulated. The sonications are thus repeated at multiple adjacent points to cover the prescribed ablation volume.

This combination of FUS-MRI has already shown convincing results on bone, prostate and uterine fibroid tumors, so the hypothesis is that it has a potential interest in the conservative treatment of breast cancer.

The Ex-Ablate 2000 system (trade name) It is a machine incorporating FUS-MRI technology. It consists of a high intensity focused ultrasound transducer mounted in the MRI examination table.

With its precision and unique ability to follow ablation, Ex-Ablate has been used in many tumor contexts and has demonstrated its ability to provide significant tumor destruction on small volumes.

On the breast, the system showed promising results in several Phase II protocols on the treatment of breast tumors with good aesthetic results and no major toxicity.

These arguments justify the choice of using Ex-Ablate as a means of thermic destruction for small size breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Woman with invasive unifocal and unilateral noninflammatory ductal breast cancer.
2. Age> 18 years.
3. Size ≤ 10 mm (measured by MRI).
4. Histological confirmation of breast cancer by biopsy with sufficient material to estimate grade, hormonal status and HER2 status.
5. Lesion well delineated in MRI after injection of gadolinium and certain ultrasound correlation with the biopsy lesion.
6. Distance> 10 mm between the tumor and the skin and between the tumor and the muscle.
7. Performance status 0 or 1
8. Biological exam according to the following standards:

   Neutrophiles> 1.5 x 109 / L Hemoglobin> 9 g / dL Plates> 100 x 109 / L ASAT - ALAT <2.5 x ULN Bilirubin <1.5 x ULN Creatinine <150 μmol / L and> 60 μmol / L Clearance> 30 ml / min
9. Informing the patient or her legal representative and signing the informed consent
10. Patient with Health care insurance available

Exclusion Criteria:

1. Invasive lobular carcinoma or extensive in-situ component or only presence of micro-calcifications as a disease sign
2. MRI or uncorrelated ultrasound lesion
3. Distance <10 mm between the tumor and the skin or nipple or chest cage or muscle
4. PS <2
5. Patient weighing more than 110 Kg
6. Breast Implants
7. History of breast irradiation
8. History of surgery on the breast to be treated (fibrous scar, staples or surgical clips)
9. Treatment with antiaromatase, tamoxifen or neoadjuvant chemotherapy within 30 days of treatment start
10. History of severe cerebrovascular disease (cerebrovascular accident within 6 months prior to inclusion) or hemolytic anemia (hematocrite <30)
11. Patient with cardiac disorders (severe hypertension, antiarrhythmic treatments, history of cardiac ischemia) 1

2. Patient under dialysis 13. Patient under anti-coagulant treatment 14. Patient refusing surgery or for which surgery is contraindicated 15. Contraindication to the realization of MRI or thermo-ablation treatment 16. Patient has a contraindication to Gadolinium 17. Vulnerable persons are defined in Article L1121-5 to -8: Pregnant women, and nursing mothers, persons deprived of their liberty by a judicial or administrative decision, persons admitted without consent under Articles L. 3212-1 and L. 3213-1 who are not covered by the provisions Of Article L. 1121-8 and persons admitted to a health or social institution for purposes other than research Persons of legal age who are under protection or who are unable to give their consent

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Histological analysis of the surgical specimen will identify the tissue destroyed by ultrasound, residual healthy tissue and possibly residual viable cancerous tissue. | up to 24 months
  All surgical specimens will be collected and analyzed in full. The sterility of the surgical specimen will be assessed using the score proposed by the EORTC-STBSG (FUS-MRI) in the local treatment of infra-centimetric breast cancer by histological confrontation of the surgical specimen

SECONDARY OUTCOMES:
Early skin toxicity is assessed until surgery | up to 24 months
  clinical examination (radiation oncologist) using NCI-CTCAE version 4.03 for erythema, telangiectasia and edema,
The quality of life will be measured before treatment on D0, and during the visit between D21 and D28 using the QLQ-C30 questionnaire - breast module BR23-version 3. | up to 24 months
  The quality of life will be measured before treatment on D0, and during the visit between D21 and D28 using the QLQ-C30 questionnaire - breast module BR23-version 3.

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTINE LOVERA, MRS, Study Director — CENTRE ANTOINE LACSSAGNE
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided